CLINICAL TRIAL: NCT05708664
Title: Precision Breast Conserving Surgery With the Guidance of Localization Combined With Multidetector CT 3-dimensional Image Reconstruction: a Single Center, Prospective, Cohort Study.
Brief Title: Precision Breast Conserving Surgery With Guidance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBCST
Record Dates: First submitted 2023-01-09; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; precision breast conserving surgery; wire-guided localization; 3-dimensional image reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PBCS (Experimental): patients enrolled in the PBCS group underwent precision breast conserving surgery guided by wire guided localization combined with MDCT guided 3D reconstruction.
  Interventions: Procedure: precision breast conserving surgery guided by wire guided localization combined with MDCT guided 3D reconstruction
- Control (No Intervention): patients enrolled in the Control group underwent palpation guided breast conserving surgery

INTERVENTIONS:
Procedure: precision breast conserving surgery guided by wire guided localization combined with MDCT guided 3D reconstruction — Local anesthesia was induced by using 1% lidocaine before wire location. The wire (localization set, PAJUNK) was placed in the superior, inferior, lateral and interior edge of the tumor through a 20-gauge needle using US guidance one day before BCS, respectively. Then, the patient underwent an immediate supine contrast enhanced CT (Philips Brilliance iCT) scan of the breast. The radiologist performed 3D reconstruction of CT images prior to surgery. Finally, the surgical procedures were performed by experienced breast surgeons combing 3D reconstruction of CT images and wire localizations one day after the localization.
  Arms: PBCS

SUMMARY:
From 2021 to 2022, 31 patients with unifocal breast cancer were enrolled for precision breast conserving surgery (PBCS) guided by wire guided localization (WGL) combined with CT guided 3D reconstruction. Surrounded WGL was performed under local anesthesia, followed by an immediate contrast enhanced CT scan. PBCS guided by CT guided 3D reconstruction was performed one day after the localization. Women who underwent palpation guided breast conserving surgery (BCS) were included as control. Two-sided Student t test, Fisher's exact test and chi-square test was applied.

DETAILED DESCRIPTION:
Background Breast conserving surgery (BCS) with radiation is accepted as a standard local treatment for early-stage breast cancer. This is largely based on the results of NSABP B-06 trial， demonstrating no significant difference in survival among patients who received total mastectomy or lumpectomy [1]. More recent studies showed that the overall survival was superior for BCS compared with mastectomy [2,3,4]. Furthermore, long-term quality of life (QoL) was better in patients treated with BCS than with mastectomy [5]. Advantages in survival and QoL have led to a higher demand for BCS.

Success of BCS is characterized by negative margins and a good cosmetic outcome. This requires doctors to precisely remove the tumor while preserving as much normal tissue as possible. Current guidelines strongly recommend achieving "no ink on tumor" for invasive breast cancer (IBC) . More widely clear margins do not significantly decrease the rate of ipsilateral breast cancer recurrence (IBCR) [6]. However, conventional localization techniques only provide approximate tumor center and fail to provide tumor extents [7]. In clinical practice, doctors may remove more tissue to achieve negative margins and avoid a reoperative intervention. Among the patients treating with BCS, 30% survivals were dissatisfied with the cosmetic outcome [8].

Wire-guided localization (WGL) is a feasible, widely used technology used for the localization of nonpalpable breast lesions prior to surgical management. The flexible self-retaining wire can be inserted into the exact lesion guided by ultrasound (US) or mammography. The surgeon than uses the wire as a guide to excise the lesion [9]. At the same time, the metal needle is visible under CT. The role of multidetector CT (MDCT) is limited in the diagnosis of breast tumors [10,11]. However, MDCT has many unique advantages. First of all, patients are in the supine position during MDCT scan, which is consistent with the surgical position. Secondly, MDCT is effective for the detection of tumor extension [12]. Beside, MDCT is convenient for 3-dimensional (3D) reconstruction. MDCT guided 3D reconstruction has been widely used in clinic, including surgery guidance. Therefore, we speculate that WGL combined with MDCT can be helpful for precision breast conserving surgery (PBCS).

The aims of this cohort study were to determine whether WGL combined with MDCT guided 3D reconstruction could guide PBCS, and to access the cosmetic outcome reported by patients.

Study Design We did a single center, prospective, cohort study in one group of our department from August 2021 to June 2022. The treatment for all patients were discussed by the multi-disciplinary team in our center. The decision in this study was decided by shared decision-making between patients and multi-disciplinary teams. All procedures for the enrolled patients were performed by one surgeon. All CT images were processed by an experienced radiologist. All specimens were evaluated by two experienced pathologists.

The study was conducted with the approval of the institutional ethics committee of The First Affiliated Hospital with Nanjing Medical University (2021-SR-226) and complied with the Declaration of Helsinki. Informed consent was obtained from all patients.

Pathologic Evaluation Pathologists performed intraoperative frozen section analysis. The size of the breast specimen was measured, and the specimen was sliced sequentially into 5mm sections. Then, the length of the margins and the size of the tumor were measured with both the naked eye and microscope. Ink on tumor was defined as a positive margin. When a positive margin was encountered, the surgeon decided to perform an additional incision or a total mastectomy. After the surgery, hematoxylin eosin stain was also performed to confirm the intraoperative analysis and the final report was subject to hematoxylin eosin stain. All pathological examinations were performed by two pathologists with more than 10 years of experience in breast pathologic examination independently.

Patient reported outcomes (PROs) Breast Cancer Treatment Outcome Scale (BCTOS) cosmetic subscale was used to access patient reported cosmetic outcomes in our study [19]. The cosmetic subscale of BCTOS contains 8 items (showing in Supplementary Table 1) designed to assess womens'subjective evaluations of cosmetic outcomes of breast cancer treatment. Each item is rated on a scale of 1 to 4 by the patient, with 1 indicated no difference compared with the untreated breast, 2 slight, 3 moderate, and 4 a large difference. The score was derived from the mean of the answers for each item, with higher scores indicating more adverse effects. Participants completed the scale at baseline (before surgery), 1 month post operation and 6 months post radiotherapy (RT). The scores were statistically analyzed to show the cosmetic changes reported by patients.

Statistical Analysis Quantitive data were reported as the mean with standard deviation. The sample size was calculated as 31 in the PBCS group. The baseline characteristics in the two groups were well balanced. So, the differences between the two groups were analyzed with the chi-square test or Fisher's exact test for categorical variables and the Student t test for continuous variables. All P values were two-sided with 5% significance levels. All analyses were performed using the software STATA version 11.0 (Computer Resource Center, America).

ELIGIBILITY:
Inclusion Criteria:

* women with T1/T2 invasive breast cancer confirmed by core biopsy
* be suitable for BCS
* the tumor should be unilateral and unifocal which is clearly visible with US

Exclusion Criteria:

* patients with an extensive intraductal component in invasive cancer
* patients who were pregnant or breast-feeding
* patients receiving neoadjuvant therapies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
The sum of located margin resection widths | 1 month post operation
  The sum of the resection widths of located superior, inferior, lateral and interior margins

SECONDARY OUTCOMES:
The specimen diameter | 1 month post operation
  The diameter of the breast specimen was measured by pathologists
the largest margin resection width | 1 month post operation
  the largest resection width of the located superior, inferior, lateral and interior margins
Operation time | intraoperative
  the duration of the surgery
Patients reported outcomes | participants completed the scale at baseline (before surgery), 1 month post operation and 6 months post radiotherapy (RT)
  Breast Cancer Treatment Outcome Scale (BCTOS) cosmetic subscale was used to access patient reported cosmetic outcomes in our study.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Xie, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Wrubel E, Natwick R, Wright GP. Breast-Conserving Therapy is Associated with Improved Survival Compared with Mastectomy for Early-Stage Breast Cancer: A Propensity Score Matched Comparison Using the National Cancer Database. Ann Surg Oncol. 2021 Feb;28(2):914-919. doi: 10.1245/s10434-020-08829-4. Epub 2020 Jul 13. PMID 32661849
- [Background] Kim H, Lee SB, Nam SJ, Lee ES, Park BW, Park HY, Lee HJ, Kim J, Chung Y, Kim HJ, Ko BS, Lee JW, Son BH, Ahn SH. Survival of Breast-Conserving Surgery Plus Radiotherapy versus Total Mastectomy in Early Breast Cancer. Ann Surg Oncol. 2021 Sep;28(9):5039-5047. doi: 10.1245/s10434-021-09591-x. Epub 2021 Jan 25. PMID 33492542
- [Background] Li P, Li L, Xiu B, Zhang L, Yang B, Chi Y, Xue J, Wu J. The Prognoses of Young Women With Breast Cancer (</=35 years) With Different Surgical Options: A Propensity Score Matching Retrospective Cohort Study. Front Oncol. 2022 Feb 28;12:795023. doi: 10.3389/fonc.2022.795023. eCollection 2022. PMID 35296009
- [Background] Hanson SE, Lei X, Roubaud MS, DeSnyder SM, Caudle AS, Shaitelman SF, Hoffman KE, Smith GL, Jagsi R, Peterson SK, Smith BD. Long-term Quality of Life in Patients With Breast Cancer After Breast Conservation vs Mastectomy and Reconstruction. JAMA Surg. 2022 Jun 1;157(6):e220631. doi: 10.1001/jamasurg.2022.0631. Epub 2022 Jun 8. PMID 35416926
- [Background] Moran MS, Schnitt SJ, Giuliano AE, Harris JR, Khan SA, Horton J, Klimberg S, Chavez-MacGregor M, Freedman G, Houssami N, Johnson PL, Morrow M; Society of Surgical Oncology; American Society for Radiation Oncology. Society of Surgical Oncology-American Society for Radiation Oncology consensus guideline on margins for breast-conserving surgery with whole-breast irradiation in stages I and II invasive breast cancer. J Clin Oncol. 2014 May 10;32(14):1507-15. doi: 10.1200/JCO.2013.53.3935. Epub 2014 Feb 10. PMID 24516019
- [Background] Leiloglou M, Kedrzycki MS, Elson DS, Leff DR. ASO Author Reflections: Towards Fluorescence Guided Tumor Identification for Precision Breast Conserving Surgery. Ann Surg Oncol. 2022 Dec;29(Suppl 3):564-565. doi: 10.1245/s10434-021-10626-6. Epub 2021 Aug 18. No abstract available. PMID 34406539
- [Background] Hill-Kayser CE, Vachani C, Hampshire MK, Di Lullo GA, Metz JM. Cosmetic outcomes and complications reported by patients having undergone breast-conserving treatment. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):839-44. doi: 10.1016/j.ijrobp.2011.08.013. Epub 2011 Dec 2. PMID 22137022
- [Background] Ahmed M, Rubio IT, Klaase JM, Douek M. Surgical treatment of nonpalpable primary invasive and in situ breast cancer. Nat Rev Clin Oncol. 2015 Nov;12(11):645-63. doi: 10.1038/nrclinonc.2015.161. Epub 2015 Sep 29. PMID 26416152
- [Background] O'Connell AM, Karellas A, Vedantham S, Kawakyu-O'Connor DT. Newer Technologies in Breast Cancer Imaging: Dedicated Cone-Beam Breast Computed Tomography. Semin Ultrasound CT MR. 2018 Feb;39(1):106-113. doi: 10.1053/j.sult.2017.09.001. Epub 2017 Sep 5. PMID 29317032
- [Background] He Z, Chen Z, Tan M, Elingarami S, Liu Y, Li T, Deng Y, He N, Li S, Fu J, Li W. A review on methods for diagnosis of breast cancer cells and tissues. Cell Prolif. 2020 Jul;53(7):e12822. doi: 10.1111/cpr.12822. Epub 2020 Jun 12. PMID 32530560
- [Background] Doihara H, Fujita T, Takabatake D, Takahashi H, Ogasawara Y, Shimizu N. Clinical significance of multidetector-row computed tomography in breast surgery. Breast J. 2006 Sep-Oct;12(5 Suppl 2):S204-9. doi: 10.1111/j.1075-122X.2006.00323.x. PMID 16959003